CLINICAL TRIAL: NCT06823947
Title: A Phase 1, Placebo-Controlled, Double-Blind, Randomized, Single and Multiple Ascending-Dose Study of KK3910 in Healthy Volunteers and Patients With Essential Hypertension
Brief Title: Study of KK3910 in Healthy Volunteers and Patients With Essential Hypertension
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 3910-001
Record Dates: First submitted 2025-02-07; First posted 2025-02-12 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteers Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- KK3910 (Experimental)
  Interventions: Drug: KK3910

INTERVENTIONS:
Drug: Placebo — Placebo is administered single dose or multiple dose by SC injection.
  Arms: Placebo
Drug: KK3910 — KK3910 is administered single dose or multiple dose by SC injection.
  Arms: KK3910

SUMMARY:
Part 1 : To evaluate the safety of single-dose KK3910 in healthy volunteers. Part 2 : To evaluate the safety of multiple-dose KK3910 in patients with essential hypertension.

ELIGIBILITY:
Inclusion Criteria: Part 1

* Voluntary consent to participate in this study must be given (in writing)
* Japanese or non-Asian healthy men 18 to < 55 years at the time of informed consent ( Japanese healthy men 65 to < 80 years for the elderly cohort)
* BMI is within the specified range at screening

Inclusion Criteria: Part 2

* Voluntary consent to participate in this study must be given (in writing)
* Japanese patients with essential hypertension, aged 18 to <65 years at the time of informed consent
* BMI is within the specified range at screening

Exclusion Criteria: Part 1

* History of any respiratory disease, heart disease, gastrointestinal disease, renal disease, liver disease, psychiatric disorder, autoimmune disease, or malignant tumor that may affect assessments in the study, as judged by principal investigator or subinvestigator.
* History of or current drug allergy
* History of or current alcoholism or drug addiction
* Smoking within the specified period
* infection within the specified period
* Any condition judged by the investigator or subinvestigator to be unsuitable for participation in the study

Exclusion Criteria: Part 2

* History of any respiratory disease, heart disease, gastrointestinal disease, renal disease, liver disease, psychiatric disorder, autoimmune disease, or malignant tumor that may affect assessments in the study, as judged by principal investigator or subinvestigator.
* History or of current drug allergy
* History of or current alcoholism or drug addiction
* Pregnant or breastfeeding patients, or patients willing to have a child during the study
* Smoking within the specified period
* infection within the specified period
* Any condition judged by the investigator or subinvestigator to be unsuitable for participation in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Part 1 : Day 1 to Day 85, Part 2: Day 1 to Day 155
  For adverse events that occurred after administration of the investigational drug, number of subjects with AEs and occurrence frequency are evaluated.

SECONDARY OUTCOMES:
Time to the maximum concentration | Part 1 : Day 1 to Day 85, Part 2 : Day 1 to Day 155
The maximum concentration | Part 1 : Day 1 to Day 85, Part 2 : Day 1 to Day 155
Area under the concentration-Time curve | Part 1 : Day 1 to Day 85, Part 2 : Day 1 to Day 155

CONTACTS AND LOCATIONS:
Overall Officials: Tatsuhiko Makine, Study Chair — Kyowa Kirin Co., Ltd.
Locations (1):
- Kitasato University Kitasato Institute Hospital, Minato-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available. The datasets generated and/or analyzed during the study sponsored by Kyowa Kirin will be available in the Vivli repository, https://vivli.org/ourmember/kyowa-kirin/ as long as conditions of data disclosure specified in the policy section of the Vivli website are satisfied.
URL: https://vivli.org/ourmember/kyowa-kirin/